CLINICAL TRIAL: NCT05094960
Title: Development of a Fast and Sensitive Method for Measurement of Circulating Cell-free DNA (cfDNA) for Diagnosis and Prognosis of Various Diseases and Evaluation of Tissue Damage Following Trauma
Brief Title: Measurement of Circulating Cell-free DNA (cfDNA) for Diagnosis and Prognosis of Various Diseases and Evaluation of Tissue Damage
Status: Completed | Type: Observational
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SOR4636CTIL
Record Dates: First submitted 2021-10-12; First posted 2021-10-26 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Correlation of cFDNA During CPB to Laboratories SIRS Parameters and Clinical Outcomes
Keywords: cfDNA-Circulating cell-free DNA; CPB-cardiopulmonary bypass; SIRS-systemic inflammatory response syndrome
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Years
Biospecimen Retention: Samples With DNA — Blood test
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood samples — 5 blood samples for each patient during CABG (coronary artery bypass grafting) surgery pre/on/post cardiopulmonary bypass machine

SUMMARY:
To characterize the changes in circulating cell-free DNA (cfDNA) levels during cardiopulmonary bypass (CPB) and to access their association with outcomes compared to standard scores.

DETAILED DESCRIPTION:
In a prospective study, the investigators enrolled seventy-one consecutive patients undergoing non-emergent coronary artery bypass grafting. Blood was drawn at baseline, after 20 and 40 minutes on CPB, after cross-clamp removal, and 30 minutes after chest closure. cfDNA was measured in sera by fluorescent method.

The investigators hypothesize that cfDNA measured by will reflect the magnitude of inflammation induced by CPB. Thus, these measurements could serve for the real-time prognosis of patients undergoing cardiac surgery. The investigators correlate cFDNA to laboratories and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Elective coronary artery bypass grafting surgery

Exclusion Criteria:

* Age < 18
* Non elective surgery
* other than CABG surgery
* Redo CABG

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult (>18yo), undergoing non-emergent first-time CABG.
Sampling Method: Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2009-07-30 (Actual); Primary Completion 2011-03-22 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
prolong LOS-length of stay | > 18 hours after the surgery
  intensive care unit length of stay
Mortality | short term - 30day; long term > 1year
  Mortality

SECONDARY OUTCOMES:
Neutrophil-NETosis | 2 hours after the surgery
  Neutrophil extracellular traps (NETs) released from activated neutrophils that undergo NETosis.

IPD SHARING:
Plan to Share IPD: No